CLINICAL TRIAL: NCT07389980
Title: Prospective Trial of the Efficacy and Safety of a Personalized Regimen of High-dose Aflibercept 8mg on Treatment-naive Polypoidal Choroidal Vasculopathy: the PALLAS Trial
Acronym: PALLAS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Min Sagong, Professor, Yeungnam University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-10-050
Record Dates: First submitted 2025-12-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Polypoidal Choroidal Vasculopathy; Polypoidal Choroidal Vasculopathy (PCV)
Keywords: PCV; Polypoidal Choroidal Vasculopathy; PALLAS; Aflibercept 8 mg
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aflibercept 8 mg (Experimental): The first loading injection will be performed for all participants. After 4 weeks, treatment response will be judged. If the polyp is completely regressed with no disease activity, injection interval will be extended to 8 weeks. The participants with presence of disease activity will continue 4-week loading injections up to 3 monthly loading dose and commence the T&E phase thereafter. In the T&E phase, patients have their injection interval extended or shortened by 4 weeks. The injection interval is maintained if the criteria for treatment adjustment were not met and residual ﬂuid was decreased from the previous visit. The minimum and maximum injection intervals are 8 and 24 weeks, respectively.
  Interventions: Drug: aflibercept 8 mg

INTERVENTIONS:
Drug: aflibercept 8 mg — The first loading injection will be performed for all participants. After 4 weeks, treatment response will be judged. If the polyp is completely regressed with no disease activity, injection interval will be extended to 8 weeks. The participants with presence of disease activity will continue 4-week loading injections up to 3 monthly loading dose and commence the T&E phase thereafter. In the T&E phase, patients have their injection interval extended or shortened by 4 weeks. The injection interval is maintained if the criteria for treatment adjustment were not met and residual ﬂuid was decreased from the previous visit. The minimum and maximum injection intervals are 8 and 24 weeks, respectively.

SUMMARY:
The purpose of this study is to evaluate the efﬁcacy and safety of the aflibercept 8 mg used in a personalized regimen, with flexible loading dose and treatment intervals from 8 to 24 weeks in eyes with treatment-naive PCV.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male or female patients ≥ 19 years of age at screening
3. Presence of active polypoidal lesions in the macular as shown by ICGA and presence of serosanguinous maculopathy (exudative or hemorrhagic features involving the macula on floor fundus photography, FA and SD-OCT AND presence of IRF or SRF that affects the central subfield as seen by SD-OCT
4. Best-corrected visual acuity (BCVA) score between 83 and 23 letters, inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts at both screening and baseline visit (study eye)

Exclusion Criteria:

1. Ocular conditions/disorders at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require planned medical or surgical intervention during the first 12-month study period, structural damage of the fovea, atrophy or fibrosis at the center of the fovea (study eye)
2. A history of any evidence of type 2 or type 3 neovascularization, myopic choroidal neovascularization, or other ocular disorders
3. Total area of subretinal hemorrhage larger than 9DA or comprising ≥ 50% of the lesion area or presence of vitreous hemorrhage in study eye
4. Any active intraocular or periocular infection or active intraocular inflammation, at screening or baseline (study eye)
5. Uncontrolled glaucoma defined as intraocular pressure (IOP) > 25 mmHg on medication, or according to investigator's judgment, at screening or baseline (study eye)
6. Ocular treatments: any anti-VEGF drugs, intraocular or periocular steroids, macular laser photocoagulation or PDT, previous ocular surgery except cataract surgery (study eye)
7. Stroke or myocardial infarction during the 6-month period prior to baseline
8. Systemic anti-VEGF therapy at any time.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-12-24 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who reached a treatment interval of ≥16 weeks at Week 96 | Week 96

SECONDARY OUTCOMES:
Last injection interval at week 96 | Week 96
Best corrected visual acuity (BCVA) at weet 96 | Week 96
  Measurement with the Early Treatment Diabetic Retinopathy Study (ETDRS) letters score
Central retinal thickness and choroidal thickness at week 96 | Week 96
  Average retinal thickness at the central 1 mm diameter
umber of participants with treatment-related adverse events | Week 96
  Slit lamp examination and fundoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided